CLINICAL TRIAL: NCT07162259
Title: Real-world Cohort Study on Sequential Therapy With ADC Drugs Following Progression of Endocrine Therapy Guided by Molecular Biomarkers in HR-positive/HER2-negative Advanced Breast Cancer
Brief Title: Cohort Study on Sequential ADC Therapy in HR-positive/HER2-negative Advanced Breast Cancer
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yan Xue (Other)
Responsible Party: Sponsor-Investigator, Yan Xue, Director of the First Department of Oncology, Xi'an International Medical Center Hospital, Xi'an International Medical Center Hospital
Organization: Xi'an International Medical Center Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025006
Record Dates: First submitted 2025-08-18; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1 (HER2 IHC 2+) (Experimental): Patients will be assigned to Cohort 1 (HER2 Immunohistochemistry，IHC，2+) based on different HER2 immunohistochemical expression levels, where they will first receive T-DXd treatment, followed by SG treatment upon disease progression.
  Interventions: Drug: First-line T-DXd followed by SG upon disease progression
- Cohort 2 (HER2 IHC ≤1+) (Experimental): Patients will be assigned to Cohort 2 (HER2 IHC ≤1+) based on different HER2 immunohistochemical expression levels, where they will first receive SG treatment, followed by T-DXd treatment upon disease progression.
  Interventions: Drug: First-line SG followed by T-DXd upon progression

INTERVENTIONS:
Drug: First-line T-DXd followed by SG upon disease progression — Patients will be assigned to Cohort 1 (HER2 IHC 2+) based on different HER2 immunohistochemical expression levels, where they will first receive T-DXd treatment, followed by SG treatment upon disease progression.
  Arms: Cohort 1 (HER2 IHC 2+)
Drug: First-line SG followed by T-DXd upon progression — Patients will be assigned to Cohort 2 (HER2 IHC ≤1+) based on different HER2 immunohistochemical expression levels, where they will first receive SG treatment, followed by T-DXd treatment upon disease progression.
  Arms: Cohort 2 (HER2 IHC ≤1+)

SUMMARY:
The combination of cyclin-dependent kinase 4/6 inhibitors (CDK4/6i) and endocrine therapy is the standard first-line treatment for advanced HR+ (hormone receptor-positive)/HER2- (human epidermal growth factor receptor 2-negative) breast cancer. However, the optimal treatment strategy after CDK4/6i progression remains unclear. In recent years, antibody-drug conjugates (ADCs) such as sacituzumab govitecan (SG) and trastuzumab deruxtecan (T-DXd) have demonstrated significant activity in HR+/HER2- breast cancer, providing new options post-CDK4/6i progression. Yet, the optimal sequencing of different ADCs (e.g., SG followed by T-DXd vs. T-DXd followed by SG) after CDK4/6i failure remains uncertain. Determining how to further optimize treatment selection to prolong survival and improve quality of life has become a key research focus in clinical practice. This study aims to explore the efficacy, safety, and potential resistance mechanisms of biomarker-guided sequential ADC therapy (e.g., SG→T-DXd vs. T-DXd→SG) following CDK4/6i progression. The findings may guide clinical decision-making and provide evidence for precision medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ≥18 years old;
2. Histologically or cytologically confirmed HR+/HER2- (HER2 IHC 0/IHC 1+ or IHC 2+ with FISH-negative) locally advanced unresectable or metastatic breast cancer, as defined by ASCO/CAP guidelines;
3. Prior treatment with CDK4/6i combined with endocrine therapy, with radiologically confirmed disease progression;
4. Presence of evaluable lesions;
5. Received ≤2 lines of chemotherapy for advanced disease;
6. Adequate organ function and performance status (ECOG score ≤2);
7. Signed informed consent.

Exclusion Criteria:

1. Previous treatment with topoisomerase 1 (TOP-1) inhibitor-based therapy;
2. Severe cardiac, hepatic, or renal dysfunction or other serious comorbidities;
3. History of moderate to severe interstitial lung disease (ILD) with concurrent pulmonary insufficiency;
4. Symptomatic brain metastases;
5. History of allergy to key components of the investigational ADC drugs (e.g., payload, antibody, or linker);
6. Patients with active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or a history of intestinal obstruction or gastrointestinal (GI) perforation;
7. Uncontrolled cardiovascular diseases (e.g., NYHA Class III/IV heart failure, myocardial infarction within 6 months);
8. Active infections (e.g., HIV, active HBV/HCV infection);
9. Pregnant or lactating women.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS1) | From the date of signing the informed consent form until the date of first documented disease progression after initial ADC therapy or date of death from any cause (whichever occurs first), assessed up to 24 months.
  PFS1 is defined as the time from signing the informed consent form to the first documented disease progression after initial ADC therapy or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression-Free Survival 2 (PFS2) | From the date of initiation of the second ADC therapy (ADC2) until the date of further documented disease progression or date of death from any cause (whichever occurs first), assessed up to 24 months.
  PFS2 is defined as the time from the initiation of the second ADC therapy (ADC2) after progression on the first ADC therapy to the date of further disease progression or death from any cause, whichever occurs first.
Composite Progression-Free Survival (PFS-Total) | From the date of signing the informed consent form until the date of the first documented disease progression (during ADC1 or ADC2 therapy) or date of death from any cause (whichever occurs first), assessed up to 36 months.
  PFS-Total is defined as the time from signing the informed consent form to the earliest occurrence of disease progression or death from any cause, regardless of whether it occurs during the first ADC therapy (ADC1), the second ADC therapy (ADC2) following progression, or thereafter.
Overall Survival (OS) | From the date of randomization until the date of death from any cause, assessed up to 60 months.
  OS is defined as the time from randomization to death due to any cause.
Objective Response Rate（ORR） | At least 4 weeks after first documented response

CONTACTS AND LOCATIONS:
Overall Officials: Yan Xue, Principal Investigator — Xi'an International Medical Center Hospital
Locations (1):
- Xi'an International Medical Center Hospital, Xi'an, China

IPD SHARING:
Plan to Share IPD: No
Since the research data involves patient privacy and intellectual property protection from collaborating institutions, the original data will not be publicly shared at this time. Summarized results will be published in academic papers.